CLINICAL TRIAL: NCT04534543
Title: MAESTRO Study: Metabolic Imaging to Improve Patient-Specific Therapy Outcomes
Acronym: MAESTRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Hanneke W. M. van Laarhoven, Head of the Department of Medical Oncology, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Volgt2
Record Dates: First submitted 2020-07-21; First posted 2020-09-01 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Gastrointestinal Cancer Metastatic
Keywords: gastrointestinal cancer; human biology; non-invasive chemistry imaging; MR imaging; spectroscopy
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: • In this study we will investigate whether biochemical imaging of change (Δ, figure 1) in the metabolic phospholipid ratios of PME and PDE between baseline and after 2 weeks of therapy are predictive for RECIST progression in gastrointestinal cancer patients after the first 9 week treatment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging (Other): Participants will undergo multiple 7T MR imaging sessions which include advanced 31P MRSI techniques, before start of palliative chemotherapy and during treatment until progression of disease or until week 54.
  Interventions: Radiation: MRI/Spectroscopy

INTERVENTIONS:
Radiation: MRI/Spectroscopy — Participants will undergo multiple 7T MR imaging sessions which include advanced 31P MRSI techniques, before start of palliative chemotherapy and during treatment until progression of disease or until week 54.

SUMMARY:
Patients suffering metastasized gastrointestinal cancer often receive ineffective treatments for prolonged periods of time as therapy non-response, which is hard to detect, cannot be determined earlier than nine weeks following start of therapy. Current therapy evaluation strategies primarily focus on morphological changes via RECIST criteria. However, morphological changes are subjected to prior physiological and metabolic alterations. Therefore, the MAESTRO project's ambition is to lay the foundations of a new area of research: the study of human biology using non-invasive chemistry imaging. For this, MAESTRO aims to unite two areas of research: metabolomics and magnetic resonance (MR). Metabolomics studies body functions through the measurements of metabolites; MR imaging (MRI) and spectroscopy (MRS) can provide 3D images of the body and measure metabolite and lipid content respectively. Previous studies show that phospholipid metabolites in particular the cell membrane precursors i.e. phosphomonoesters (PME), and the cell membrane degradation products i.e. phosphodiesters (PDE) are valuable biomarkers in therapy assessment. With this MAESTRO approach, the consortium aims at reducing the nine weeks period before therapy efficacy evaluation to three weeks or less. By validating the powerful new MRS(I)-visible biomarkers in a patient cohort, a non-invasive technology can be developed for dynamically mapping biochemical processes in the whole human body and pave the way for individualized medicine.

DETAILED DESCRIPTION:
Primary objective

-In this study we will investigate whether biochemical imaging of change (Δ, figure 1) in the metabolic phospholipid ratios of PME and PDE between baseline and after 2 weeks of therapy are predictive for progression free survival (PFS) and/or overall survival (OS) in gastro-oesophageal cancer patients within 27 weeks of treatment.

Secondary objectives:

* In this study we will investigate whether biochemical imaging of change (Δ, figure 1) in the metabolic phospholipid ratios of PME and PDE between baseline and after 2 weeks of therapy are predictive for RECIST progression in gastro-oesophageal cancer patients after the first 9 week treatment period.
* Investigate whether biochemical imaging of the metabolic phospholipid ratios of PME and PDE at baseline of therapy are predictive for RECIST progression after the first 9-week treatment period, and for PFS and OS in gastro-oesophageal cancer patients.
* Investigate whether biochemical imaging of change (δ, figure 1) in the metabolic phospholipid ratios of PME and PDE after a 9-week treatment period are predictive for RECIST progression following that treatment period, and for PFS and OS in gastro-oesophageal cancer patients.
* Exploratory multi variable analysis for the development of a prediction model to predict resistance to treatment within 3 weeks after the start of chemotherapy with the use of all chemistry imaging data including all MR detectable nuclei and clinical parameters.

Study population: We aim to include a total of 70 patients with metastatic gastro-oesophageal cancer before start of palliative chemotherapy.

Intervention: Participants will undergo multiple 7T MR imaging sessions which include advanced 31P MRSI techniques, before start of palliative chemotherapy and during treatment until progression of disease or until week 9.

Main study parameters/endpoints: Study parameters include; metabolic ratios of the phospholipids PME and PDE from the area under the curve (AUC) of the corresponding spectral peaks, size measurements from CT and MRI scans, coded radiology reports, clinical patient data, e.g. chemotherapy details extracted from clinical notes which are coded before storage to preserve anonymity. Main endpoint is defined by progression or death after 27 weeks measured using the RECIST progression criteria for which chemical imaging its predictive value is investigated in the primary objective.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: Patients will be asked for three extra hospital visits to undergo 7T MRI of approximately one hour per session (3x 1 hour). MRI is a safe non-invasive technique without use of ionizing radiation and so far, extensive research has not shown any side-effects of the high magnetic field used in 7T MRI, resulting in low inherent risks for the participants. This study will be started only after approval of the IGJ and the medical device investigation agency of the AMC. Patients' therapy is not delayed by participation in this study and patients with MRI contraindications are excluded from participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver metastasis of gastrointestinal cancer, with histological or cytological proof of metastasis or a high suspicion on CT imaging.
* Tumour size ≥ 1cm.
* WHO-performance score 0-2.
* Scheduled for first- or second-line palliative chemotherapy containing capecitabine combined with oxaliplatin (CAPOX) or fluorouracil combined with oxaliplatin and folinic acid (FOLFOX).
* Written informed consent.

Exclusion Criteria:

* Any psychological, familial, sociological, or geographical condition potentially hampering adequate informed consent or compliance with the study protocol.
* Contra-indications for MR scanning, including patients with a pacemaker, cochlear implant or neurostimulator; patients with non-MR compatible metallic implants in their eye, spine, thorax or abdomen; or a non-MR compatible aneurysm clip in their brain; patients with claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
PME/PDE-ratio from Area Under the Curve (AUC): predictive | 72 months
  The primary outcome measure in this study is the PME/PDE-ratio (PME/PDE) resulting from the AUC of the metabolite peaks in the acquired metabolic images e.g. spectra.
  This measure is used to calculate changes in the metabolic phospholipid-ratios of PME and PDE (ΔPME/PDE) between baseline and after 2 weeks of therapy. In addition, this outcome measure is used to investigate secondary objectives including PME/PDE at baseline as a sole predictor (see Outcome Measure 3).
Change in PME/PDE (ΔPME/PDE): predictive | 72 months
  The second primary outcome measure to investigate the discriminative ability of PME/PDE is the ΔPME/PDE between baseline and after 2 weeks of therapy.
  This measure is used to investigate the primary objective whether biochemical imaging of change in the metabolic phospholipid-ratios of PME and PDE (ΔPME/PDE) between baseline and after 2 weeks of therapy are predictive for RECIST progression in gastrointestinal cancer patients after the first 9 week treatment period. In addition, this outcome measure is also used to investigate secondary objectives which includes different time periods over which ΔPME/PDE is measured.

SECONDARY OUTCOMES:
PME/PDE at baseline: predictive | 72 months
  This secondary measure is used investigate the secondary objective whether biochemical imaging of PME/PDE at baseline of therapy is predictive for RECIST progression after the first 9-week treatment period, and for PFS and OS in gastrointestinal cancer patients. PME/PDE at baseline results from the AUC of the metabolite peaks in the acquired metabolic images e.g. specta (see also Outcome Measure 1).
Prediction model | 72 months
  Exploratory multi variable analysis for the development of a prediction model to predict resistance to treatment within 3 weeks after the start of chemotherapy with the use of all chemistry imaging data including all MR detectable nuclei and clinical parameters.
  Multi-variable analysis of clinically relevant data to investigate the feasibility of a dynamic prediction model will use all chemical imaging data, size measurements from CT, conventional 7T MR imaging scans, coded radiology reports, clinical patient data, e.g. chemotherapy details extracted from clinical notes which are coded before storage to preserve anonymity, choice of therapy, progression free survival (PFS) and overall survival (OS) and metastasis origin.
(Δ)PME/PDE predictive significance | 72 months
  To investigate to what extent baseline PME/PDE and (ΔPME/PDE) over all different time periods is predictive of PFS and OS, we will use standard survival analysis techniques (e.g. Cox regression, accelerated failure time models) and estimate the C-index as measure of discriminative ability.
Response to treatment | 72 months
  This outcome measure results from conventional therapy evaluation defined by RECIST progression. It is used in the primary and secondary objectives as the gold standard for the therapy evaluation predictors assessed in this study (ΔPME/PDE, PME/PDE, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke WM van Laarhoven, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - UMC Utrecht, Utrecht